CLINICAL TRIAL: NCT04661995
Title: Notched Noise Therapy for Suppression of Tinnitus: A Randomized Controlled Trial
Brief Title: Notched Noise Therapy for Suppression of Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C3281-W; 1IK2RX003281-01A2 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-12-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Tinnitus; Notched Noise Therapy
Keywords: Tinnitus; Notched Noise Therapy
MeSH Terms: conditions — Tinnitus | interventions — Hearing Aids; NADP Transhydrogenases

STUDY DESIGN:
Intervention Model Description: A formal randomized controlled trial assessing Amplification + Notched-Noise Therapy (NNT), Amplification + Broadband Noise (BBN), or Amplification-Only (A-O) as treatments for tinnitus will be conducted. 108 participants will be tested on four occasions: baseline, and 4, 8, and 12 weeks post-baseline. Sound delivery for all participants will be accomplished using hearing aids to stream the custom notched noise filter software to the device. These participants will use the devices during most/all waking hours for 8 weeks and will be blinded to the type of stimulus they are receiving. Participants in all three groups will complete outcome measures at week 0 (baseline), week 4 (first in-course assessment), and week 8 (final in-course assessment). Treatment will be discontinued after 8 weeks, with a follow-up assessment at 12 weeks.
Who Masked: Participant
Masking Description: Participants in all three groups will be blinded to the randomization of tinnitus treatment. Three treatment groups are identified: Amplification + Notched Noise Therapy; Amplification + Broadband Noise (white noise); and Amplification Only. Participants will be blinded to the treatment they are receiving so that results of perceptual change of subjective tinnitus can be truly measured with validated, evidence-based outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Amplification + Notched Noise Therapy (Experimental): Following the baseline assessment, participants will be randomly assigned to one of the study groups. This treatment group will include a Notched Noise Therapy, a 1-10 kHz noise "notched" within a 1-octave range centered around the psychoacoustic tinnitus pitch match measured. Randomized participants will wear their hearing aids with this loaded software for 8 weeks. They will be seen at a baseline, 4 week, and 8 week visits for outcome measures and any adjustments in hearing aid comfort.
  Interventions: Combination Product: Hearing Aid and Notched Noise Therapy
- Amplification + Broadband Noise (Active Comparator): Following the baseline assessment, participants will be randomly assigned to one of the study groups. A popular and commonly used sound therapy treatment, this treatment group will listen to a broadband noise, or "white noise," that is housed on the manufacturer's hearing aid tinnitus program. They will be seen at a baseline, 4 week, and 8 week visits for outcome measures and any adjustments in hearing aid comfort.
  Interventions: Combination Product: Hearing Aid and Broadband Noise
- Amplification Only (Placebo Comparator): Following the baseline assessment, participants will be randomly assigned to one of the study groups. Hearing aids are ear-level, self-contained, FDA-approved hearing device. Hearing aids help individuals with hearing loss and provide safe amplification/gain to frequencies that have loss.
  Interventions: Device: Hearing Aid

INTERVENTIONS:
Combination Product: Hearing Aid and Notched Noise Therapy — Notched Noise Therapy involves presenting wide-band sound with the tinnitus frequency region notched out, referred to as notched noise, or notch therapy. This procedure may distribute lateral inhibition into the notched frequency region, suppressing tinnitus neural activity believed to be occurring there. This type of therapy is provided through a sound file that is streamed through hearing aids.
  Other Names: HA + NNT
  Arms: Amplification + Notched Noise Therapy
Combination Product: Hearing Aid and Broadband Noise — Broadband Noise, or "white noise," is a common tinnitus sound therapy treatment option. It is also commonly used as a "masker" noise for individuals with tinnitus that like to enrich their environment with sound.
  Other Names: HA + BBN
  Arms: Amplification + Broadband Noise
Device: Hearing Aid — A-O groups will use ear-level, self-contained devices (hearing aids) that (1) are capable of streaming shapeable broadband noise between 1-10 kHz; (2) allow for normal conversation; and (3) are comfortable, easy to use, and discrete. These criteria describe a behind-the-ear hearing aid with the capability of streaming custom sounds. Hearing aids are used to provide amplification to those with hearing loss and are fit by licensed audiologists. Sometimes, hearing aids can provide benefit to those with bothersome tinnitus.
  Other Names: A-O
  Arms: Amplification Only

SUMMARY:
Tinnitus ("ringing in the ears") has long been a problem for Veterans. The problem continues to escalate due to high levels of noise in the military, and because tinnitus often is associated with traumatic brain injury and post-traumatic stress disorder. In spite of limited research support, sound-based (acoustic) therapies are most often used for tinnitus intervention, and increasing numbers of commercial devices are becoming available that offer various acoustic-stimulus protocols. The proposed study will provide evidence from a randomized controlled trial comparing effects of acoustic-stimulus methods that are purported to suppress tinnitus and/or reduce its functional effects. The study will focus on methods with the strongest scientific rationale, i.e., noise that is notched around the predominant tinnitus-frequency region. Special ear-level devices will deliver these acoustic-therapy protocols that are purported to modify tinnitus-related neural activity. The study will follow a study recently completed by the applicant that provides preliminary evidence supporting this method.

DETAILED DESCRIPTION:
Tinnitus is the most prevalent service-connected disability for Veterans. Many Veterans are offered sound-based (acoustic) therapy for tinnitus that is intended to alter the tinnitus perception and/or reactions to tinnitus in a clinically beneficial way. Various methods of acoustic therapy are in use and companies are promoting different products. It remains unknown; however, how certain acoustic parameters may be more effective than others. Recent research has shown the benefit of one such acoustic therapy, Notched Noise Therapy, that presents wideband sound with the tinnitus frequency region notched out, theorized to distribute lateral inhibition into the notched frequency region to suppress neural activity believed to cause the tinnitus percept. Previous studies have typically involved brief daily exposures, which are not as likely to remodel neural processes underlying tinnitus as is continuous "immersion" in background sound, which is adopted here. The proposed study will conduct a randomized controlled trial to evaluate the efficacy of notched noise therapy (NNT). The long-term goal of the research program is to develop an accessible, evidence-based treatment that reduces tinnitus loudness and to be able to assess that treatment through a validated method of behavioral and physiological clinical tools. The overall objective for this CDA-2 research plan, which is the next step toward attainment of the investigators' long-term goal, is to systematically evaluate the utility of functional, psychoacoustic, and electrophysiologic measures to reveal the overall whole-health impact in Veterans with chronic tinnitus. The trial will enroll 108 participants, who will be randomized to one of three acoustic therapy methods: amplification + notched noise, amplification + noise without notch, and amplification-only. The three groups will be asked to wear ear-level devices (combination instruments that provide both amplification and 1-10 kHz shapeable noise) as much as possible during waking hours. All participants will undergo acoustic therapy for 8 weeks and will complete outcome measures (i.e., Tinnitus Functional Index, Psychoacoustic loudness and pitch matches, AEP, and EEG measures) at baseline and at 4 and 8 weeks. They will repeat outcome assessment at 12 weeks to evaluate for maintenance of any effects while not receiving acoustic therapy for 4 weeks. (Participants requiring hearing aids for hearing loss will continue to use their aids during the 4-week no-treatment period). The investigators hypothesize that NNT suppresses tinnitus perception by distributing lateral inhibition into the notched frequency region and will therefore, reduce the perception of tinnitus loudness. At the completion of this CDA-2 program, the expected outcomes include a NNT as a therapy for tinnitus and the contributions that it may have on tinnitus perception as well as a solid training foundation for a successful VA research career. These results are expected to have an important positive impact because they will not only provide insight into the true reactionary and perceptual benefit of an intervention, but a treatment evaluation protocol will be determined, ultimately providing a foundation for the development of evidence-based acoustic therapies to treat tinnitus, a critical component and goal of Veteran tinnitus care.

ELIGIBILITY:
Inclusion Criteria:

Candidates must meet the following inclusion criteria to qualify:

* Veteran
* no active middle-ear disease
* at least one air conduction hearing threshold of 40 dB HL or worse in each ear between .25-8 kHz as measured at the first study visit
* unilateral or bilateral constant tinnitus
* index score on the Tinnitus Functional Index (TFI) of at least 25 (out of a maximum score of 100)
* a score of 24 or higher on the Mini Mental State Exam (MMSE)
* a tinnitus pitch match between 2-10 kHz (and achieve desired level of precision as described below in 3.3 Study Procedures, Tinnitus Psychoacoustic Assessment)
* demonstrates understanding of the requirements of the study
* motivated and capable of participating (including ability to communicate in English)

Exclusion Criteria:

The following exclusion criteria will be used:

* two or more hearing thresholds exceeding 70 dB HL
* significant conductive hearing loss-defined as an air-bone gap of 15 dB at more than two frequencies in one ear, or an air-bone gap greater than 15 dB at any one frequency
* suspicion of secondary (somatic) tinnitus, Meniere's disease, or tinnitus potentially related to temporo-mandibular disorder or whiplash (any of which can be ruled out with an examination by an appropriate physician)
* any mental, emotional, or health conditions that would preclude full study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of Tinnitus Functional Index Scores from Baseline at 4 weeks, 8 weeks, and 12 weeks | 4 time points/visits: Baseline, 4 weeks, 8 weeks, 12 weeks
  The TFI is useful in both clinical and research settings because of its excellent responsiveness to treatment-related change, its high construct validity for scaling the overall severity of tinnitus, and its comprehensive coverage of the negative impacts of tinnitus (Meikle, et al., 2012; Henry, Griest et al., 2016). Participants will complete the TFI at each appointment prior to any audiometric or psychoacoustic testing.

SECONDARY OUTCOMES:
Change of Tinnitus Loudness Match from Baseline at 4 weeks, 8 weeks, and 12 weeks | 4 time points/visits: Baseline, 4 weeks, 8 weeks, 12 weeks
  For tinnitus loudness match, participants will be seated facing a computer monitor and shown how to use the TES Module (device with a knob and four buttons) to respond to acoustic signals presented through Etymotic ER-4B insert earphones. Test frequencies include 0.25-16 kHz in 1/3-octave intervals. Participants will complete the Tinnitus Loudness Match at each appointment to identify change in loudness perception.

OTHER OUTCOMES:
Change of Electroencephalography (EEG) power in delta, theta, alpha, beta, and gamma bands from Baseline to 8 weeks | 2 time points/visits: Baseline, 8 weeks
  30 participants (10 from each study arm) will be randomized into a supplemental group to receive extra testing: EEG assessment. EEG will be recorded using an Electro-Cap International, Inc. cap housing 64 Ag/AgCl electrodes and the Neuroscan recording system. Responses from all 64 electrode channels will be available for analysis, thus allowing for identification of channels with the strongest responses. Data will be re-sampled to 128 Hz, band-pass filtered to 2-44 Hz and subsequently transposed, plotted, and carefully inspected for manual artifact rejection and epochs containing excessive artifacts will be removed. Average Fourier cross-spectral matrices will be computed for bands delta (2-3.9 Hz), theta (4-7.9 Hz), alpha1 (8-9.9 Hz), alpha 2 (10-12.9 Hz), beta1 (13-18.4 Hz), beta2 (18.5-21.4 Hz), beta3 (21.5-30.4 Hz), and gamma (30.5-44 Hz).
Change of N100, P200, and P300 Auditory Evoked Potentials (AEPs) from Baseline to 8 weeks | 2 time points/visits: Baseline, 8 weeks
  Two different AEP protocols will be used to assess neural activity associated with auditory attention in this subset of study participants (10 from each arm) at two timepoints: baseline and after 8 weeks of amplification with or without additional sound therapy. AEPs will be recorded using an Electro-Cap International, Inc. cap housing 64 Ag/AgCl electrodes and the Neuroscan recording system. The two AEP protocols are: (1) A paired-click P50 paradigm will be used to assess auditory habituation, which is part of the process of sensory gating. (2) An auditory P300 paradigm will be used to assess higher-level attentional mechanisms. Stimuli will include 500 Hz pure tones (frequent stimulus) and 1000 Hz pure tones (rare stimulus). During this protocol, AEP components N100, P200, and P300 will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Candice Manning Quinn, PhD AuD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No